CLINICAL TRIAL: NCT04020614
Title: Assessment of Colorectal Cancer Awareness in Patients Admitted to the General Surgery Outpatient Clinic
Brief Title: Colorectal Cancer Awareness in Turkey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Collaborators: Istanbul Training and Researh Hospital (Unknown); Taksim Training and Research Hospital (Unknown)
Responsible Party: Principal Investigator, Cemile Idiz, Principal Investigator, Istanbul University
Other Study IDs: Colorectal Cancer
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Awareness; Screening
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survey: All of the patients that enrolled in this study will be in this group.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — A survey with 13 questions will be applied to the patients

SUMMARY:
Colorectal cancer is among the most common types of cancer worldwide. Population-based screening programs for breast, cervical, and colorectal cancer have been introduced as part of cancer control in many high-income countries. Population-based cancer screening programs do not exist in most low- and middle-income countries. There are some studies that report the awareness of colorectal cancer in Turkey.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common type of cancer in both men and women. According to World Health Organization data, in 2012, 694 thousand people were thought to be due to colorectal cancer and this number increased to 862 thousand people in 2018. Especially in most low- and middle-income countries where cancers are mainly detected through very-late-stage symptoms and many are not reported. Recent researches may lead to new approaches to early detection and treatment using improved awareness of the symptomatic disease and population-based screening of asymptomatic people. The increasing of colorectal cancer awareness could help early detection of colorectal cancers. In this study, the investigators aimed to determine the level of awareness of colorectal cancer and knowledge about colorectal cancer screenings in patients who applied to general surgery outpatients clinic where a colorectal cancer diagnosis was most frequently diagnosed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who apply to the general surgery outpatients clinic

Exclusion Criteria:

* Younger than 18 years old
* Older than 80 years old
* Mental retardation or other mental illness
* Refusing to join the study

Ages: 18 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients who apply to the general surgery outpatient clinic with any diseases.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-08-15 (Estimated)

PRIMARY OUTCOMES:
The awareness of patients about colorectal cancer | 3 months
  To assess the awareness of patients about colorectal cancer with a survey

CONTACTS AND LOCATIONS:
Overall Officials: Coskun Cakir, MD, Study Director — Istanbul Training and Research Hospital
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
In case of request individual participant data could be shared with other researchers

REFERENCES:
- [Result] Andsoy II, Gul A. Breast, cervix and colorectal cancer knowledge among nurses in Turkey. Asian Pac J Cancer Prev. 2014;15(5):2267-72. doi: 10.7314/apjcp.2014.15.5.2267. PMID 24716968
- [Result] Kaya O, Hoca O, Kulacoglu H. Knowledge and awareness of auxiliary health personnel about colorectal cancer. Turk J Gastroenterol. 2013;24(4):339-44. doi: 10.4318/tjg.2013.0631. PMID 24254266